CLINICAL TRIAL: NCT00603564
Title: A Comparison of CPAP Delivered by Helmet and O2 Therapy With Venturi Mask for the Treatment of Acute Respiratory Failure in Community-acquired Pneumonia
Brief Title: Helmet Continuous Positive Airway Pressure Versus Oxygen Venturi in Acute Respiratory Failure in CAP: CAPOVeRSO
Acronym: CAPOVeRSO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely interrupted because patients randomized to CPAP reached the endpoint quicker than anticipated in the protocol
Sponsor: University of Milan (Other)
Responsible Party: Roberto Cosentini, MD, Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPOVeRSO 01
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-10

CONDITIONS: Pneumonia; Community-Acquired Infections; Respiratory Insufficiency; Acute Lung Injury
Keywords: CPAP; community-acquired pneumonia; acute respiratory failure; hypoxemia; Continuous Positive Airway Pressure
MeSH Terms: conditions — Pneumonia; Community-Acquired Infections; Respiratory Insufficiency; Acute Lung Injury; Community-Acquired Pneumonia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): CPAP delivered by a helmet
  Interventions: Procedure: Castar Starmed (CPAP) delivered by a helmet
- 2 (No Intervention): O2 administration via a conventional Venturi mask

INTERVENTIONS:
Procedure: Castar Starmed (CPAP) delivered by a helmet — Continuous Positive Airway Pressure delivered by a helmet with PEEP valve of 10 cmH2O and FiO2 0.5
  Other Names: Castar Starmed CP209/2
  Arms: 1

SUMMARY:
The purpose of this study is to compare the efficacy of CPAP application by a helmet and O2 administration by a Venturi mask in terms of gas exchanges improvement in patients with acute respiratory failure due to community-acquired pneumonia.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is one of the commonest causes of hospitalised acute respiratory failure with a mortality rate up t 30%.

Continuous Positive Airway Pressure (CPAP) has ben recently proved to be effective. To date, however, no prospective randomised study has been published on the comparison between CPAP and O2 administration via a Venturi mask for the treatment of acute respiratory failure in immunocompetent patients with community-acquired pneumonia.

Therefore, the aim of this study is to compare the efficacy of CPAP delivered by a helmet and O2 administration via a Venturi mask in terms of gas exchanges improvement in early acute respiratory failure (PaO2/FiO2 between 210 and 285)due to community-acquired pneumonia.

A Steering Committee composed by the principal investigators will request an interim analysis at 20% enrolment in order to monitor the criteria for equipoise of the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Community-acquired pneumonia (CAP) defined as: new chest x-ray pulmonary infiltrate, fever, and respiratory symptoms
* Acute Hypoxemic Respiratory failure
* Respiratory Rate < 35 breaths/min
* PaO2/FiO2 > 200 and < 300 while breathing oxygen for at least 15 minutes via a Venturi mask with FiO2 0.5

Exclusion criteria

* Immunosuppression
* acute cardiogenic pulmonary edema
* Patients belonging to Class II-III-IV of the NYHA
* Acute coronary syndrome
* Acute Respiratory Acidosis pH < 7.35 and PaCO2 > 45 mmHg
* More than 3 acute organ failures
* Systolic Pressure < 90 mmHg under fluid resuscitation or vasopressor drug use
* Seizures
* Decreased level of consciousness (GCS <12)
* Inability to clear secretions
* Pre-defined intubation criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: roberto cosentini, MD, Study Chair — Ospedale Maggiore Policlinico Mangiagalli e Regina Elena
Locations (1):
- Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan, Italy

REFERENCES:
- [Background] Gregg RW, Friedman BC, Williams JF, McGrath BJ, Zimmerman JE. Continuous positive airway pressure by face mask in Pneumocystis carinii pneumonia. Crit Care Med. 1990 Jan;18(1):21-4. doi: 10.1097/00003246-199001000-00006. PMID 2403506
- [Background] Hilbert G, Gruson D, Vargas F, Valentino R, Chene G, Boiron JM, Pigneux A, Reiffers J, Gbikpi-Benissan G, Cardinaud JP. Noninvasive continuous positive airway pressure in neutropenic patients with acute respiratory failure requiring intensive care unit admission. Crit Care Med. 2000 Sep;28(9):3185-90. doi: 10.1097/00003246-200009000-00012. PMID 11008980
- [Derived] Cosentini R, Brambilla AM, Aliberti S, Bignamini A, Nava S, Maffei A, Martinotti R, Tarsia P, Monzani V, Pelosi P. Helmet continuous positive airway pressure vs oxygen therapy to improve oxygenation in community-acquired pneumonia: a randomized, controlled trial. Chest. 2010 Jul;138(1):114-20. doi: 10.1378/chest.09-2290. Epub 2010 Feb 12. PMID 20154071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Steering Committee requested an interim analysis at 20% enrollment in order to monitor the criteria for actual equipoise of the two treatments. Being this unplanned, the Lan-DeMets approach was followed and a manifest superiority of the CPAP treatment was identified, with a nominal alpha exceeding the criterion for interruption set at 0.00008.
Groups:
- CPAP (Continuous Positive Airway Pressure): CPAP delivered by a helmet
- Venturi: O2 administration via a conventional Venturi mask
Period: Overall Study
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Venturi
Started | 20 (January 2006) | 27 (January 2006)
Completed | 20 (February 2008) | 27 (February 2008)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Venturi | Total
Number analyzed (Participants) | 20 | 27 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 12 | 19 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (17) | 72 (13) | 69 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach an Improvement in Terms of Gas Exchange, Defined as a PaO2/FiO2 Ratio ≥315
Time Frame: on admission and at 1, 6, 12, 24 and 48 hours until PaO2/FiO2 ratio ≥315
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Venturi
Number analyzed (Participants) | 20 | 27
minute | 405 (855) | 2437 (1170)
Statistical Analysis 1: Comparison: CPAP (Continuous Positive Airway Pressure) vs Venturi; endpoint was analyzed in terms of time by comparison of mean +- SD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: PaO2/FiO2 Ratio Mantainance
Description: the number of subjects who could maintain, once reached, a PaO2/FiO2 ratio ≥315 at 1 and 24 hours after the qualifying measurement
Time Frame: 1, 6, 12, 24 and 48 hours
Measure: Number; unit: participants
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Venturi
Number analyzed (Participants) | 20 | 27
participants | 19 | 8
Statistical Analysis 1: Comparison: CPAP (Continuous Positive Airway Pressure) vs Venturi; Test type: Superiority or Other; p = 0.000007, Chi-squared

ADVERSE EVENTS:
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Venturi
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/27
Other Adverse Events (participants affected / at risk) | 0/20 | 0/27

LIMITATIONS AND CAVEATS:
Limitations of our study are mainly related to the early reaching of the end-point of the CPAP group. We were not able to evaluate the safety of the CPAP application and to address conclusions on its efficacy on outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No